CLINICAL TRIAL: NCT00043186
Title: A Randomized, Double-Blind, Placebo-controlled, Multi-dose Phase 2 Study to Determine the Efficacy, Safety and Tolerability of AMG 162 in the Treatment of Postmenopausal Women With Low Bone Mineral Density
Brief Title: Determine the Efficacy, Safety and Tolerability of Denosumab (AMG 162) in the Treatment of Postmenopausal Women With Low Bone Mineral Density
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20010223
Record Dates: First submitted 2002-08-06; First posted 2002-08-07 (Estimated); Results first posted 2010-07-28 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Low Bone Mineral Density
Keywords: bone loss; osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Denosumab; Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (9):
- Placebo (Placebo Comparator): Participants received double-blind subcutaneous (SC) placebo injections every 3 months until month 21 and then placebo SC injections once every 6 months from Month 24 through Month 42.
  Interventions: Drug: Placebo
- Denosumab 6 mg every 3 months (Experimental): Participants received denosumab 6 mg SC every 3 months until Month 21 and then denosumab 60 mg every 6 months from Month 24 through Month 42.
  Interventions: Drug: Denosumab
- Denosumab 14 mg every 3 months (Experimental): Participants received denosumab 14 mg SC every 3 months until Month 21 and then denosumab 60 mg every 6 months from Month 24 through Month 42.
  Interventions: Drug: Denosumab
- Denosumab 30 mg every 3 months (Experimental): Participants received denosumab 30 mg SC every 3 months until Month 21 then placebo SC every 6 months at Month 24 and Month 30 and then denosumab 60 mg SC every 6 months at Month 36 and Month 42.
  Interventions: Drug: Denosumab
- Denosumab 14 mg every 6 months (Experimental): Participants received denosumab 14 mg SC every 6 months until Month 21 and then denosumab 60 mg every 6 months from Month 24 through Month 42.
  Interventions: Drug: Denosumab
- Denosumab 60 mg every 6 months (Experimental): Participants received denosumab 60 mg SC every 6 months until Month 42.
  Interventions: Drug: Denosumab
- Denosumab 100 mg every 6 months (Experimental): Participants received denosumab 100 mg SC every 6 months until Month 21 and then denosumab 60 mg every 6 months from Month 24 through Month 42.
  Interventions: Drug: Denosumab
- Denosumab 210 mg every 6 months (Experimental): Participants received denosumab 210 mg SC every 6 months until Month 21 and then placebo every 6 months from Month 24 through Month 42.
  Interventions: Drug: Denosumab
- Alendronate 70 mg (Active Comparator): Participants received open-label alendronate 70 mg tablets orally once a week through Month 24. From Month 24 to Month 48 participants received no treatment.
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Placebo — Placebo subcutaneous injection
  Arms: Placebo
Drug: Denosumab — Denosumab for subcutaneous injection
  Other Names: AMG 162; Prolia
  Arms: Denosumab 100 mg every 6 months; Denosumab 14 mg every 3 months; Denosumab 14 mg every 6 months; Denosumab 210 mg every 6 months; Denosumab 30 mg every 3 months; Denosumab 6 mg every 3 months; Denosumab 60 mg every 6 months
Drug: Alendronate — Alendronate 70 mg tablets
  Other Names: Fosamax
  Arms: Alendronate 70 mg

SUMMARY:
To determine the effect of denosumab treatment compared with placebo over 12 months on bone mineral density (BMD) of the lumbar spine in postmenopausal women with low BMD. The clinical hypothesis is that denosumab subcutaneous injections administered every 3 or 6 months for 12 months will significantly increase lumbar spine bone mineral density and will be well tolerated.

ELIGIBILITY:
Inclusion Criteria

* women not more than 80 years of age on date of randomization
* ≥ 1 year postmenopausal on date of randomization
* ambulatory
* if ≤ 60 years of age, or had or would require a bilateral oophorectomy, serum follicle stimulating hormone (FSH) > 50 mU/mL or serum estradiol < 20 pg/mL
* low BMD (BMD T-score ≤ -1.8 at any 1 of the following sites: lumbar spine, femoral neck, or total hip; BMD T-scores must not have been < -4.0 at the lumbar spine or - 3.5 at the femoral neck or total hip)
* before any study-specific procedure, including the screening dual X-ray absorptiometry (DXA) scan, gave informed consent for participation in the study.

Exclusion Criteria

* fluoride treatment for osteoporosis within the 2 years before the enrollment date
* bisphosphonate use within the 12 months before the enrollment date
* administration of the following medications within the 6 months before the enrollment date

  * tibolone
  * Parathyroid hormone (PTH) (or any derivative)
  * systemic glucocorticosteroids (> 5 mg oral prednisone equivalent per day for > 10 days)
  * inhaled corticosteroids (> 2000 μg per day for > 10 days)
  * anabolic steroids or testosterone
* administration of the following medications within the 3 months before the enrollment date

  * systemic hormone replacement therapy
  * selective estrogen receptor modulators
  * calcitonin
  * calcitriol
* current hyper- or hypothyroidism (allowed if stable on thyroid replacement therapy and thyroid-stimulating hormone was within the normal range)
* current hyper- or hypoparathyroidism
* albumin-adjusted serum calcium < 8.5 mg/dL (< 2.125 mol/L)
* osteomalacia
* rheumatoid arthritis
* Paget's disease
* malignancy within the 5 years before enrollment (except cervical carcinoma in situ or basal cell carcinoma, which were acceptable)
* renal disease; ie, creatinine clearance ≤ 35 mL/min
* any bone disease, other than osteoporosis, which could interfere with the interpretation of the findings (eg, osteogenesis imperfecta or osteopetrosis)
* malabsorption syndrome
* weight, height, or girth that could preclude accurate DXA measurements
* < 2 lumbar vertebrae (L1 through L4) evaluable by DXA
* recent long bone fracture (within 6 months)
* osteoporotic-related fracture (ie, crush or wedge vertebral fracture or hip fracture) known or suspected to have occurred within 2 years of randomization
* > 1 single, grade 1 vertebral fracture
* currently enrolled in or had participated within the previous 30 days in other investigational device or drug trial(s) (For some trials, this may have been allowed after discussion and written approval from Amgen.)
* known sensitivity to mammalian-derived drug preparations (eg, Herceptin®)
* any organic or psychiatric disorder, serum chemistry, or hematology that, in the opinion of the investigator, could have prevented the subject from completing the study or have interfered with the interpretation of the study results
* self-reported alcohol or drug abuse within the previous 12 months
* any disorder that compromised the ability to give truly informed consent for participation in the study
* previous administration of denosumab
* known sensitivity or contraindication to alendronate
* known sensitivity or contraindication to tetracycline derivatives (subjects in the biopsy substudy only).

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2002-05; Primary Completion 2007-04 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Beck TJ, Lewiecki EM, Miller PD, Felsenberg D, Liu Y, Ding B, Libanati C. Effects of denosumab on the geometry of the proximal femur in postmenopausal women in comparison with alendronate. J Clin Densitom. 2008 Jul-Sep;11(3):351-9. doi: 10.1016/j.jocd.2008.04.001. Epub 2008 May 20. PMID 18495508
- [Result] Lewiecki EM, Miller PD, McClung MR, Cohen SB, Bolognese MA, Liu Y, Wang A, Siddhanti S, Fitzpatrick LA; AMG 162 Bone Loss Study Group. Two-year treatment with denosumab (AMG 162) in a randomized phase 2 study of postmenopausal women with low BMD. J Bone Miner Res. 2007 Dec;22(12):1832-41. doi: 10.1359/jbmr.070809. PMID 17708711
- [Result] McClung MR, Lewiecki EM, Cohen SB, Bolognese MA, Woodson GC, Moffett AH, Peacock M, Miller PD, Lederman SN, Chesnut CH, Lain D, Kivitz AJ, Holloway DL, Zhang C, Peterson MC, Bekker PJ; AMG 162 Bone Loss Study Group. Denosumab in postmenopausal women with low bone mineral density. N Engl J Med. 2006 Feb 23;354(8):821-31. doi: 10.1056/NEJMoa044459. PMID 16495394
- [Result] Miller PD, Bolognese MA, Lewiecki EM, McClung MR, Ding B, Austin M, Liu Y, San Martin J. Effect of denosumab on bone density and turnover in postmenopausal women with low bone mass after long-term continued, discontinued, and restarting of therapy: a randomized blinded phase 2 clinical trial. Bone. 2008 Aug;43(2):222-229. doi: 10.1016/j.bone.2008.04.007. Epub 2008 Apr 26. PMID 18539106
- [Result] Peterson MC, Riggs MM. A physiologically based mathematical model of integrated calcium homeostasis and bone remodeling. Bone. 2010 Jan;46(1):49-63. doi: 10.1016/j.bone.2009.08.053. Epub 2009 Sep 2. PMID 19732857
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject Enrolled: 11-May-2002 Last Subject Enrolled: 30-Apr-2003
Groups:
- Denosumab 6 mg Q3M: Participants received denosumab 6 mg SC every 3 months (Q3M) until Month 21 and then denosumab 60 mg every 6 months from Month 24 through Month 42.
- Denosumab 14 mg Q3M: Participants received denosumab 14 mg SC every 3 months until Month 21 and then denosumab 60 mg every 6 months from Month 24 through Month 42.
- Denosumab 30 mg Q3M: Participants received denosumab 30 mg SC every 3 months until Month 21 then placebo SC every 6 months at Month 24 and Month 30 and then denosumab 60 mg SC every 6 months at Month 36 and Month 42.
- Denosumab 14 mg Q6M: Participants received denosumab 14 mg SC every 6 months (Q6M) until Month 21 and then denosumab 60 mg every 6 months from Month 24 through Month 42.
- Denosumab 60 mg Q6M: Participants received denosumab 60 mg SC every 6 months until Month 42.
- Denosumab 100 mg Q6M: Participants received denosumab 100 mg SC every 6 months until Month 21 and then denosumab 60 mg every 6 months from Month 24 through Month 42.
- Denosumab 210 mg Q6M: Participants received denosumab 210 mg SC every 6 months until Month 21 and then placebo every 6 months from Month 24 through Month 42.
Period: Overall Study
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Started | 46 | 44 | 44 | 41 | 54 | 47 | 42 | 47 | 47
Completed | 29 | 29 | 24 | 19 | 36 | 39 | 25 | 31 | 30
Not Completed | 17 | 15 | 20 | 22 | 18 | 8 | 17 | 16 | 17
Not completed — Physician Decision | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 2 | 2 | 2 | 3 | 2 | 1 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 11 | 8 | 11 | 13 | 14 | 6 | 12 | 9 | 10
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Disease progression | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 4 | 0
Not completed — Ineligibility determined | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 3 | 5 | 1 | 1 | 1 | 1 | 1 | 1 | 2
Not completed — Noncompliance | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg | Total
Number analyzed (Participants) | 46 | 44 | 44 | 41 | 54 | 47 | 42 | 47 | 47 | 412
Age Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (9.1) | 62.8 (8.6) | 62.3 (6) | 61.2 (8.5) | 61.4 (8.1) | 63.1 (8.1) | 64.9 (8.2) | 60.5 (7.8) | 62.8 (8.2) | 62.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 44 | 44 | 41 | 54 | 47 | 42 | 47 | 47 | 412
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 37 | 33 | 42 | 36 | 49 | 39 | 37 | 42 | 40 | 355
  Black or African American | 0 | 1 | 1 | 2 | 1 | 1 | 3 | 0 | 3 | 12
  Hispanic or Latino | 8 | 8 | 1 | 3 | 3 | 5 | 2 | 5 | 4 | 39
  Asian | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4
  Japanese | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 12 for the Placebo and Denosumab Arms
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry. Percent change from Baseline to Month 12 calculated using ((Month 12 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and Month 12
Population: Randomized participants with non-missing Baseline and non-missing value at Month 12.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M
Number analyzed (Participants) | 40 | 36 | 36 | 32 | 48 | 41 | 37 | 41
Percent change | -0.81 (0.48) | 4.41 (0.50) | 4.71 (0.50) | 6.69 (0.54) | 3.03 (0.43) | 4.55 (0.47) | 5.52 (0.49) | 5.07 (0.47)
Statistical Analysis 1: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.87, 95% CI [4.59 to 7.16]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.33, 95% CI [5.01 to 7.65]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.35, 95% CI [4.07 to 6.64]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.84, 95% CI [2.60 to 5.07]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 7.50, 95% CI [6.13 to 8.87]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.52, 95% CI [4.19 to 6.85]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.21, 95% CI [3.88 to 6.55]

2. Secondary Outcome: Serum CTX Percent Change From Baseline at Month 12
Description: Serum C-Telopeptide (CTX). Percent change from Baseline to Month 12 calculated using ((Month 12 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and Month 12
Population: Randomized participants with non-missing Baseline and non-missing value at Month 12
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 36 | 35 | 36 | 31 | 47 | 41 | 36 | 42 | 40
Percent change | -4.699 [-20.74 to 28.3] | -61.366 [-74.42 to -41.92] | -77.989 [-87.02 to -55.37] | -87.238 [-90.53 to -71.25] | -12.054 [-38.48 to 10.69] | -70.757 [-81.47 to -55.78] | -78.617 [-85.85 to -60.95] | -84.107 [-90.70 to -77.85] | -72.603 [-81.72 to -59.55]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.166, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Urine NTX/Creatinine Percent Change From Baseline at Month 12
Description: Urinary N-telopeptide (uNTX)/Creatinine. Percent change from Baseline to Month 12 calculated using ((Month 12 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and Month 12
Population: Randomized participants with non-missing Baseline and non-missing value at Month 12.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 36 | 35 | 36 | 31 | 47 | 40 | 36 | 42 | 40
Percent change | 24.300 [-23.06 to 39.84] | -40.018 [-49.76 to -6.38] | -54.688 [-66.80 to -23.33] | -60.652 [-73.16 to -46.40] | -2.027 [-20.30 to 10.84] | -36.523 [-54.67 to -16.06] | -51.256 [-67.31 to -22.17] | -58.502 [-70.55 to -29.84] | -45.409 [-59.96 to -22.74]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.020, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 12 for the Alendronate Arm
Description: as for outcome 1
Time Frame: Baseline and Month 12
Population: Randomized participants with non-missing Baseline and non-missing value at Month 12.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alendronate 70 mg
Number analyzed (Participants) | 45
Percent change | 4.59 (0.45)

5. Secondary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 24
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry. Percent change from Baseline to Month 24 calculated using ((Month 24 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 24 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 24.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 34 | 32 | 33 | 27 | 41 | 41 | 33 | 36 | 39
Percent change | -1.25 (0.68) | 7.42 (0.69) | 7.21 (0.68) | 8.83 (0.76) | 3.94 (0.60) | 7.19 (0.62) | 7.31 (0.67) | 7.86 (0.65) | 6.09 (0.63)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 7.34, 95% CI [5.56 to 9.12]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 9.11, 95% CI [7.31 to 10.91]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 8.56, 95% CI [6.71 to 10.41]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 8.44, 95% CI [6.69 to 10.19]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.19, 95% CI [3.43 to 6.94]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 10.08, 95% CI [8.14 to 12.01]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 8.46, 95% CI [6.62 to 10.30]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 8.66, 95% CI [6.80 to 10.53]

6. Secondary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 36
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry. Percent change from Baseline to Month 36 calculated using ((Month 36 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 36 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 36.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 30 | 31 | 25 | 23 | 38 | 38 | 29 | 38 | 33
Percent change | -1.80 (0.82) | 8.57 (0.80) | 9.17 (0.89) | 1.94 (0.94) | 7.99 (0.72) | 9.04 (0.74) | 10.63 (0.82) | 0.85 (0.72) | 4.70 (0.78)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.50, 95% CI [4.32 to 8.67]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.013, ANCOVA; Mean Difference (Final Values) = 2.65, 95% CI [0.55 to 4.75]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 12.43, 95% CI [10.19 to 14.68]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 10.84, 95% CI [8.74 to 12.94]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 9.79, 95% CI [7.69 to 11.89]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.74, 95% CI [1.37 to 6.12]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 10.97, 95% CI [8.63 to 13.32]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 10.37, 95% CI [8.16 to 12.59]

7. Secondary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 42
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry. Percent change from Baseline to Month 42 calculated using ((Month 42 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 42 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 42.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 8 | 5 | 7 | 5 | 15 | 12 | 6 | 7 | 10
Percent change | 1.09 (1.70) | 7.21 (2.13) | 10.04 (1.86) | 5.06 (2.13) | 9.46 (1.24) | 9.59 (1.40) | 9.99 (1.93) | 1.06 (1.80) | 6.51 (1.51)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.02, ANCOVA; Mean Difference (Final Values) = 5.42, 95% CI [0.89 to 9.95]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.992, ANCOVA; Mean Difference (Final Values) = -0.03, 95% CI [-5.07 to 5.02]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = 8.90, 95% CI [3.72 to 14.09]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = 8.50, 95% CI [4.15 to 12.86]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = 8.37, 95% CI [4.11 to 12.63]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.292, ANCOVA; Mean Difference (Final Values) = 3.98, 95% CI [-1.42 to 9.37]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = 8.95, 95% CI [3.94 to 13.96]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.094, ANCOVA; Mean Difference (Final Values) = 6.12, 95% CI [0.57 to 11.67]

8. Secondary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 48
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry. Percent change from Baseline to Month 48 calculated using ((Month 48 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 48 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 48.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 29 | 29 | 24 | 20 | 37 | 39 | 27 | 30 | 31
Percent change | -2.39 (1.11) | 9.35 (1.09) | 9.93 (1.20) | 9.03 (1.33) | 10.10 (0.96) | 10.34 (0.96) | 11.76 (1.13) | 2.50 (1.07) | 4.54 (1.06)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.93, 95% CI [3.97 to 9.89]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.89, 95% CI [1.92 to 7.85]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 14.15, 95% CI [11.08 to 17.21]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 12.73, 95% CI [9.94 to 15.52]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 12.49, 95% CI [9.66 to 15.32]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 11.42, 95% CI [8.12 to 14.73]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 12.32, 95% CI [9.15 to 15.49]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 11.74, 95% CI [8.72 to 14.76]

9. Secondary Outcome: Serum CTX Percent Change From Baseline at Month 24
Description: Serum C-Telopeptide (CTX). Percent change from Baseline to Month 24 calculated using ((Month 24 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 24 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 24.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 32 | 30 | 32 | 25 | 38 | 39 | 31 | 33 | 38
Percent change | -5.940 [-23.22 to 20.61] | -50.687 [-73.73 to -27.21] | -74.078 [-84.96 to -52.32] | -83.985 [-89.66 to -74.02] | -8.467 [-24.02 to 25.84] | -68.437 [-81.80 to -44.39] | -80.460 [-89.31 to -43.68] | -85.680 [-90.94 to -78.32] | -69.386 [-79.82 to -52.04]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.622, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Serum CTX Percent Change From Baseline at Month 36
Description: Serum C-Telopeptide (CTX). Percent change from Baseline to Month 36 calculated using ((Month 36 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 36 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 36.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 29 | 30 | 24 | 22 | 31 | 36 | 27 | 36 | 32
Percent change | -16.577 [-28.96 to -0.29] | -62.298 [-81.94 to -42.09] | -53.643 [-82.23 to -34.04] | 56.286 [21.35 to 73.85] | -57.500 [-75.77 to -23.56] | -54.418 [-72.02 to -12.53] | -45.057 [-81.69 to -11.29] | 72.135 [34.18 to 136.00] | -33.982 [-56.86 to -21.93]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.011, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.026, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Serum CTX Percent Change From Baseline at Month 42
Description: Serum C-Telopeptide (CTX). Percent change from Baseline to Month 42 calculated using ((Month 42 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 42 months
Population: Randomized participantswith non-missing Baseline and non-missing value at Month 42.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 23 | 27 | 21 | 16 | 30 | 35 | 24 | 31 | 27
Percent change | -16.279 [-31.66 to 18.31] | -63.543 [-83.99 to -38.15] | -40.827 [-85.17 to -13.72] | -62.334 [-88.37 to -27.85] | -46.408 [-80.65 to -32.46] | -57.255 [-74.60 to -23.04] | -56.377 [-77.35 to -20.98] | 33.999 [0.15 to 49.68] | -46.743 [-58.94 to -26.14]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.012, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.012, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.012, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.012, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Serum CTX Percent Change From Baseline at Month 48
Description: Serum C-Telopeptide (CTX). Percent change from Baseline to Month 48 calculated using ((Month 48 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 48 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 48.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 27 | 29 | 24 | 16 | 34 | 37 | 24 | 30 | 29
Percent change | -14.561 [-33.09 to 6.61] | -40.016 [-80.76 to 0.11] | -34.999 [-78.25 to -7.84] | -52.656 [-78.86 to -5.25] | -39.899 [-73.80 to -9.78] | -51.494 [-78.57 to -14.62] | -36.480 [-70.12 to -18.54] | 7.067 [-17.06 to 31.25] | -43.724 [-56.28 to -14.07]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.015, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.050, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.029, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.032, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.050, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.050, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.073, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Urine NTX/Creatinine Percent Change From Baseline at Month 24
Description: Urinary N-telopeptide (uNTX)/Creatinine. Percent change from Baseline to Month 24 calculated using ((Month 24 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 24 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 24.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 32 | 30 | 32 | 25 | 38 | 39 | 31 | 33 | 39
Percent change | 14.422 [-5.30 to 56.37] | -19.699 [-51.71 to 1.61] | -37.691 [-60.65 to -4.19] | -49.907 [-68.26 to -20.43] | 2.134 [-15.60 to 45.10] | -32.303 [-54.06 to 15.35] | -37.001 [-72.15 to 11.74] | -47.105 [-76.14 to -24.75] | -44.482 [-59.46 to -8.98]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.409, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Urine NTX/Creatinine Percent Change From Baseline at Month 36
Description: Urinary N-telopeptide (uNTX)/Creatinine. Percent change from Baseline to Month 36 calculated using ((Month 36 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 36 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 36.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 29 | 30 | 24 | 22 | 31 | 36 | 26 | 36 | 31
Percent change | 0.508 [-21.60 to 11.89] | -33.294 [-56.03 to -3.63] | -47.752 [-58.74 to -16.01] | 82.910 [32.79 to 108.70] | -44.301 [-58.12 to -15.68] | -36.874 [-57.37 to -5.32] | -27.174 [-56.30 to 25.52] | 70.997 [24.80 to 125.90] | -15.627 [-40.75 to 15.42]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.011, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.077, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Urine NTX/Creatinine Percent Change From Baseline at Month 42
Description: Urinary N-telopeptide (uNTX)/Creatinine. Percent change from Baseline to Month 42 calculated using ((Month 42 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 42 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 42.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 24 | 27 | 21 | 16 | 30 | 35 | 24 | 31 | 27
Percent change | -18.102 [-31.05 to 30.83] | -40.741 [-60.82 to -12.95] | -40.043 [-65.63 to -9.12] | -58.893 [-67.49 to -14.26] | -47.188 [-69.64 to -25.46] | -39.269 [-64.25 to -4.97] | -46.674 [-63.98 to -9.33] | 26.277 [-16.99 to 88.12] | -33.102 [-53.10 to -19.07]
Statistical Analysis 1: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.053, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.053, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.022, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.032, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.053, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.053, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.020, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.053, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Urine NTX/Creatinine Percent Change From Baseline at Month 48
Description: Urinary N-telopeptide (uNTX)/Creatinine. Percent change from Baseline to Month 48 calculated using ((Month 48 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 48 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 48.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 27 | 28 | 24 | 16 | 32 | 35 | 24 | 30 | 28
Percent change | -21.064 [-36.94 to 32.77] | -23.311 [-62.33 to 11.43] | -38.002 [-67.11 to -15.91] | -50.864 [-80.48 to -9.49] | -46.128 [-64.44 to -14.07] | -40.375 [-70.06 to -0.46] | -41.998 [-70.45 to -6.62] | 7.884 [-35.02 to 72.97] | -32.198 [-59.36 to 6.68]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.010, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.172, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.029, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.047, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.015, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.168, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.168, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.172, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 12
Description: as for outcome 1
Time Frame: Baseline and 12 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 12.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 40 | 36 | 36 | 32 | 48 | 42 | 37 | 41 | 45
Percent change | -0.56 (0.37) | 2.89 (0.38) | 2.45 (0.39) | 3.32 (0.42) | 1.94 (0.33) | 3.56 (0.36) | 2.53 (0.38) | 2.33 (0.36) | 2.11 (0.35)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 2.67, 95% CI [1.70 to 3.64]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 2.90, 95% CI [1.90 to 3.89]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.09, 95% CI [2.07 to 4.11]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.12, 95% CI [3.13 to 5.11]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 2.5, 95% CI [1.55 to 3.46]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.89, 95% CI [2.83 to 4.95]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.01, 95% CI [1.99 to 4.04]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.46, 95% CI [2.43 to 4.48]

18. Secondary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 24
Description: as for outcome 5
Time Frame: Baseline and 24 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 24.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 35 | 32 | 33 | 27 | 41 | 41 | 33 | 35 | 39
Percent change | -1.92 (0.44) | 4.04 (0.45) | 3.55 (0.44) | 5.03 (0.50) | 2.62 (0.39) | 4.96 (0.40) | 3.67 (0.44) | 4.18 (0.43) | 3.27 (0.41)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.19, 95% CI [4.04 to 6.34]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.10, 95% CI [4.93 to 7.27]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.59, 95% CI [4.40 to 6.78]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.89, 95% CI [5.76 to 8.01]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.54, 95% CI [3.41 to 5.67]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.95, 95% CI [5.69 to 8.21]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.48, 95% CI [4.29 to 6.67]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.97, 95% CI [4.76 to 7.17]

19. Secondary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 36
Description: as for outcome 6
Time Frame: Baseline and 36 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 36.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 30 | 31 | 25 | 23 | 38 | 37 | 29 | 38 | 33
Percent change | -2.84 (0.60) | 4.79 (0.58) | 4.41 (0.65) | -1.23 (0.68) | 4.31 (0.52) | 5.83 (0.54) | 4.33 (0.60) | -1.43 (0.53) | 0.93 (0.57)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.78, 95% CI [2.19 to 5.36]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.07, ANCOVA; Mean Difference (Final Values) = 1.41, 95% CI [-0.12 to 2.94]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 7.17, 95% CI [5.54 to 8.80]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 8.67, 95% CI [7.13 to 10.21]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 7.15, 95% CI [5.62 to 8.69]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.07, ANCOVA; Mean Difference (Final Values) = 1.61, 95% CI [-0.12 to 3.35]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 7.26, 95% CI [5.56 to 8.95]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 7.63, 95% CI [6.02 to 9.24]

20. Secondary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 42
Description: as for outcome 7
Time Frame: Baseline and 42 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 42.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 8 | 5 | 7 | 5 | 15 | 12 | 6 | 7 | 10
Percent change | -1.96 (1.16) | 5.01 (1.43) | 3.98 (1.28) | 2.37 (1.46) | 4.54 (0.85) | 6.34 (0.98) | 4.70 (1.32) | -2.67 (1.23) | 2.98 (1.03)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = 4.94, 95% CI [1.86 to 8.02]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.677, ANCOVA; Mean Difference (Final Values) = -0.71, 95% CI [-4.10 to 2.68]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = 6.66, 95% CI [3.14 to 10.18]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 8.29, 95% CI [5.26 to 11.33]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.50, 95% CI [3.59 to 9.41]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.047, ANCOVA; Mean Difference (Final Values) = 4.33, 95% CI [0.61 to 8.05]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Final Values) = 5.94, 95% CI [2.53 to 9.36]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = 6.97, 95% CI [3.28 to 10.66]

21. Secondary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 48
Description: as for outcome 8
Time Frame: Baseline and 48 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 48.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 29 | 29 | 24 | 20 | 37 | 39 | 27 | 30 | 31
Percent change | -3.52 (0.65) | 5.45 (0.63) | 4.03 (0.70) | 3.86 (0.77) | 4.82 (0.56) | 6.06 (0.56) | 4.99 (0.66) | -1.37 (0.62) | 1.17 (0.62)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.69, 95% CI [2.97 to 6.41]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.015, ANCOVA; Mean Difference (Final Values) = 2.16, 95% CI [0.43 to 3.89]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 8.52, 95% CI [6.74 to 10.30]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 9.58, 95% CI [7.95 to 11.21]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 8.34, 95% CI [6.70 to 9.99]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 7.38, 95% CI [5.45 to 9.31]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 7.55, 95% CI [5.72 to 9.38]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 8.97, 95% CI [7.23 to 10.72]

22. Secondary Outcome: Distal 1/3 Radius Bone Mineral Density Percent Change From Baseline at Month 12
Description: as for outcome 1
Time Frame: Baseline and 12 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 12.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 39 | 35 | 35 | 32 | 44 | 43 | 37 | 37 | 42
Percent change | -1.97 (0.50) | 0.89 (0.52) | 0.40 (0.53) | 1.10 (0.55) | 0.94 (0.46) | 1.29 (0.48) | 1.07 (0.50) | 1.09 (0.51) | -0.53 (0.47)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.033, ANCOVA; Mean Difference (Final Values) = 1.44, 95% CI [0.11 to 2.76]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.06, 95% CI [1.69 to 4.42]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.04, 95% CI [1.68 to 4.40]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.26, 95% CI [1.94 to 4.57]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 2.91, 95% CI [1.60 to 4.21]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.07, 95% CI [1.65 to 4.49]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 2.37, 95% CI [0.99 to 3.76]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 2.86, 95% CI [1.47 to 4.24]

23. Secondary Outcome: Distal 1/3 Radius Bone Mineral Density Percent Change From Baseline at Month 24
Description: as for outcome 5
Time Frame: Baseline and 24 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 24.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 34 | 32 | 32 | 27 | 38 | 41 | 33 | 33 | 35
Percent change | -2.78 (0.56) | 1.31 (0.57) | 0.62 (0.58) | 1.30 (0.63) | 2.48 (0.52) | 1.89 (0.51) | 1.48 (0.56) | 0.81 (0.56) | -0.78 (0.55)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.009, ANCOVA; Mean Difference (Final Values) = 1.99, 95% CI [0.49 to 3.49]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.58, 95% CI [2.06 to 5.10]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.26, 95% CI [2.73 to 5.78]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.09, 95% CI [2.55 to 5.62]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.67, 95% CI [3.23 to 6.11]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.26, 95% CI [3.78 to 6.73]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.08, 95% CI [2.48 to 5.68]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.39, 95% CI [1.86 to 4.93]

24. Secondary Outcome: Distal 1/3 Radius Bone Mineral Density Percent Change From Baseline at Month 36
Description: as for outcome 6
Time Frame: Baseline and 36 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 36.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 29 | 31 | 24 | 23 | 37 | 39 | 29 | 35 | 30
Percent change | -3.64 (0.63) | 1.99 (0.60) | 1.06 (0.69) | 1.05 (0.71) | 2.08 (0.55) | 2.69 (0.55) | 1.92 (0.62) | 0.12 (0.57) | -0.95 (0.61)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = 2.69, 95% CI [1.01 to 4.38]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.77, 95% CI [2.14 to 5.39]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.56, 95% CI [3.87 to 7.26]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.33, 95% CI [4.75 to 7.92]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.73, 95% CI [4.12 to 7.33]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.70, 95% CI [2.89 to 6.50]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.70, 95% CI [2.92 to 6.49]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.63, 95% CI [3.96 to 7.30]

25. Secondary Outcome: Distal 1/3 Radius Bone Mineral Density Percent Change From Baseline at Month 42
Description: as for outcome 7
Time Frame: Baseline and 42 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 42.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 3 | 1 | 3 | 1
Percent change | -6.59 (3.00) | 1.00 (3.26) | 0.82 (2.92) | -3.91 (3.39) | 1.29 (2.14) | -0.87 (2.93) | 0.02 (5.00) | 0.59 (2.52) | -3.32 (3.95)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.496, ANCOVA; Mean Difference (Final Values) = 3.27, 95% CI [-7.16 to 13.7]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.527, ANCOVA; Mean Difference (Final Values) = 6.60, 95% CI [-6.38 to 19.59]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.503, ANCOVA; Mean Difference (Final Values) = 5.72, 95% CI [-2.90 to 14.33]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.527, ANCOVA; Mean Difference (Final Values) = 2.68, 95% CI [-6.54 to 11.89]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.503, ANCOVA; Mean Difference (Final Values) = 7.41, 95% CI [-2.19 to 17.01]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.503, ANCOVA; Mean Difference (Final Values) = 7.59, 95% CI [-1.85 to 17.03]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.503, ANCOVA; Mean Difference (Final Values) = 7.18, 95% CI [-2.45 to 16.81]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.233, ANCOVA; Mean Difference (Final Values) = 7.88, 95% CI [0.78 to 14.97]

26. Secondary Outcome: Distal 1/3 Radius Bone Mineral Density Percent Change From Baseline at Month 48
Description: as for outcome 8
Time Frame: Baseline and 48 months
Population: Randomized participants with non-missing baseline and non-missing value at Month 48.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 28 | 29 | 22 | 19 | 35 | 38 | 27 | 28 | 28
Percent change | -4.67 (0.75) | 1.04 (0.73) | 1.42 (0.84) | 1.77 (0.91) | 1.74 (0.66) | 1.71 (0.65) | 1.37 (0.75) | -0.94 (0.74) | -2.67 (0.75)
Statistical Analysis 1: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.41, 95% CI [4.48 to 8.34]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.44, 95% CI [4.19 to 8.70]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.09, 95% CI [3.91 to 8.26]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.72, 95% CI [3.70 to 7.73]
Statistical Analysis 5: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.054, ANCOVA; Mean Difference (Final Values) = 2.00, 95% CI [-0.04 to 4.04]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.74, 95% CI [1.71 to 5.77]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.05, 95% CI [4.00 to 8.10]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.39, 95% CI [4.49 to 8.28]

27. Secondary Outcome: Total Body Bone Mineral Density Percent Change From Baseline at Month 12
Description: as for outcome 1
Time Frame: Baseline and 12 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 12.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 36 | 36 | 35 | 29 | 43 | 42 | 34 | 38 | 39
Percent change | -0.21 (0.46) | 1.82 (0.45) | 1.80 (0.46) | 2.74 (0.51) | 0.55 (0.41) | 2.51 (0.43) | 1.78 (0.46) | 2.08 (0.44) | 1.51 (0.44)
Statistical Analysis 1: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = 2.30, 95% CI [1.09 to 3.51]
Statistical Analysis 2: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.005, ANCOVA; Mean Difference (Final Values) = 1.73, 95% CI [0.52 to 2.93]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = 2.00, 95% CI [0.74 to 3.25]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 2.72, 95% CI [1.54 to 3.91]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.202, ANCOVA; Mean Difference (Final Values) = 0.77, 95% CI [-0.41 to 1.95]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 2.95, 95% CI [1.65 to 4.26]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = 2.02, 95% CI [0.78 to 3.26]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = 2.03, 95% CI [0.80 to 3.27]

28. Secondary Outcome: Total Body Bone Mineral Density Percent Change From Baseline at Month 24
Description: as for outcome 5
Time Frame: Baseline and 24 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 24.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 33 | 31 | 33 | 24 | 37 | 40 | 32 | 32 | 34
Percent change | -1.64 (0.53) | 2.59 (0.54) | 2.91 (0.53) | 4.44 (0.62) | 0.89 (0.49) | 2.57 (0.49) | 3.00 (0.53) | 2.75 (0.53) | 1.50 (0.52)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.14, 95% CI [1.71 to 4.56]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.40, 95% CI [2.95 to 5.84]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.64, 95% CI [3.19 to 6.09]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.22, 95% CI [2.85 to 5.58]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 2.53, 95% CI [1.13 to 3.94]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.09, 95% CI [4.53 to 7.64]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.55, 95% CI [3.12 to 5.98]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.23, 95% CI [2.76 to 5.69]

29. Secondary Outcome: Total Body Bone Mineral Density Percent Change From Baseline at Month 36
Description: as for outcome 6
Time Frame: Baseline and 36 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 36.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 28 | 31 | 25 | 21 | 35 | 39 | 27 | 36 | 28
Percent change | -1.61 (0.94) | 3.14 (0.88) | 3.04 (0.98) | 2.34 (1.09) | 2.04 (0.83) | 2.80 (0.80) | 2.59 (0.94) | -0.29 (0.83) | 4.55 (0.94)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.16, 95% CI [3.63 to 8.68]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.275, ANCOVA; Mean Difference (Final Values) = 1.32, 95% CI [-1.06 to 3.7]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.005, ANCOVA; Mean Difference (Final Values) = 4.20, 95% CI [1.65 to 6.75]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = 4.41, 95% CI [2.07 to 6.75]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.009, ANCOVA; Mean Difference (Final Values) = 3.65, 95% CI [1.25 to 6.05]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.009, ANCOVA; Mean Difference (Final Values) = 3.95, 95% CI [1.22 to 6.68]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Final Values) = 4.65, 95% CI [2.05 to 7.24]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = 4.75, 95% CI [2.28 to 7.22]

30. Secondary Outcome: Total Body Bone Mineral Density Percent Change From Baseline at Month 42
Description: as for outcome 7
Time Frame: Baseline and 42 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 42.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 6 | 2 | 1 | 3 | 1
Percent change | 1.61 (1.76) | 1.90 (3.71) | 4.05 (1.70) | 8.85 (3.07) | 3.72 (1.97) | 4.92 (1.83) | 3.79 (3.63) | -0.75 (1.50) | 2.85 (2.67)
Statistical Analysis 1: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.949, ANCOVA; Mean Difference (Final Values) = 2.18, 95% CI [-8.73 to 13.10]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.949, ANCOVA; Mean Difference (Final Values) = 3.30, 95% CI [-2.70 to 9.31]
Statistical Analysis 3: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.709, ANCOVA; Mean Difference (Final Values) = 1.24, 95% CI [-6.81 to 9.29]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.949, ANCOVA; Mean Difference (Final Values) = -2.36, 95% CI [-8.55 to 3.83]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.949, ANCOVA; Mean Difference (Final Values) = 2.10, 95% CI [-4.51 to 8.72]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.484, ANCOVA; Mean Difference (Final Values) = 7.23, 95% CI [-0.83 to 15.3]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.949, ANCOVA; Mean Difference (Final Values) = 2.44, 95% CI [-3.77 to 8.66]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.949, ANCOVA; Mean Difference (Final Values) = 0.29, 95% CI [-10.82 to 11.40]

31. Secondary Outcome: Total Body Bone Mineral Density Percent Change From Baseline at Month 48
Description: as for outcome 8
Time Frame: Baseline and 48 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 48.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 28 | 28 | 23 | 17 | 35 | 38 | 25 | 29 | 27
Percent change | -2.54 (0.99) | 3.68 (0.98) | 3.38 (1.07) | 3.76 (1.27) | 3.42 (0.86) | 3.43 (0.87) | 3.68 (1.03) | -0.29 (0.96) | 4.49 (1.00)
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 7.02, 95% CI [4.35 to 9.69]
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.092, ANCOVA; Mean Difference (Final Values) = 2.25, 95% CI [-0.37 to 4.87]
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.22, 95% CI [3.50 to 8.94]
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.97, 95% CI [3.51 to 8.43]
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.96, 95% CI [3.44 to 8.48]
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.29, 95% CI [3.25 to 9.34]
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.91, 95% CI [3.13 to 8.70]
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 6.22, 95% CI [3.58 to 8.87]

32. Secondary Outcome: Bone Specific Alkaline Phosphatase Percent Change From Baseline at Month 12
Description: Bone specific alkaline phosphatase (BSAP). Percent change from Baseline to Month 12 calculated using ((Month 12 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 12 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 12.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 36 | 35 | 36 | 31 | 47 | 40 | 36 | 42 | 39
Percent change | -4.609 [-26.46 to 30.31] | -62.716 [-77.57 to -47.64] | -60.098 [-76.61 to -41.34] | -70.256 [-80.58 to -55.16] | -39.474 [-64.97 to -13.73] | -65.215 [-77.11 to -51.79] | -61.979 [-74.25 to -50.61] | -67.634 [-75.90 to -50.19] | -61.059 [-69.89 to -46.08]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

33. Secondary Outcome: Bone Specific Alkaline Phosphatase Percent Change From Baseline at Month 24
Description: Bone specific alkaline phosphatase (BSAP). Percent change from Baseline to Month 24 calculated using ((Month 24 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 24 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 24.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 32 | 30 | 32 | 25 | 38 | 37 | 31 | 33 | 39
Percent change | 16.464 [-20.18 to 52.94] | -41.225 [-65.61 to -22.04] | -47.597 [-69.11 to -16.28] | -57.905 [-66.41 to -22.36] | -22.350 [-44.05 to 0.50] | -43.448 [-62.70 to -18.28] | -50.176 [-64.82 to -23.14] | -48.833 [-71.34 to -27.38] | -48.778 [-58.87 to -25.77]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

34. Secondary Outcome: Bone Specific Alkaline Phosphatase Percent Change From Baseline at Month 36
Description: Bone specific alkaline phosphatase (BSAP). Percent change from Baseline to Month 36 calculated using ((Month 36 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 36 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 36.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 29 | 29 | 24 | 22 | 31 | 36 | 26 | 34 | 31
Percent change | 1.955 [-28.21 to 45.67] | -39.012 [-66.11 to -12.10] | -56.021 [-69.45 to -21.31] | 22.343 [-0.27 to 49.28] | -47.500 [-63.87 to -32.19] | -42.541 [-64.46 to -24.35] | -47.418 [-57.70 to -22.78] | 61.747 [14.65 to 101.28] | -8.209 [-40.84 to 7.80]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.049, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.146, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

35. Secondary Outcome: Bone Specific Alkaline Phosphatase Percent Change From Baseline at Month 42
Description: Bone specific alkaline phosphatase (BSAP). Percent change from Baseline to Month 42 calculated using ((Month 42 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 42 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 42.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 24 | 27 | 21 | 16 | 31 | 35 | 23 | 31 | 27
Percent change | 1.288 [-25.01 to 51.68] | -40.182 [-65.62 to -11.21] | -40.819 [-64.78 to -6.13] | -52.684 [-67.62 to -34.69] | -53.763 [-62.49 to -28.55] | -44.892 [-62.36 to -25.45] | -48.303 [-59.51 to -18.60] | 17.841 [4.18 to 82.99] | -22.069 [-41.00 to 8.92]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.061, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.058, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

36. Secondary Outcome: Bone Specific Alkaline Phosphatase Percent Change From Baseline at Month 48
Description: Bone specific alkaline phosphatase (BSAP). Percent change from Baseline to Month 48 calculated using ((Month 48 value - Baseline value) / Baseline value ) x 100.
Time Frame: Baseline and 48 months
Population: Randomized participants with non-missing Baseline and non-missing value at Month 48.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Number analyzed (Participants) | 27 | 29 | 24 | 16 | 34 | 37 | 24 | 30 | 29
Percent change | 18.122 [-28.72 to 59.58] | -34.727 [-56.34 to 3.83] | -45.779 [-60.49 to 9.42] | -47.770 [-60.61 to -30.76] | -46.286 [-57.67 to -24.26] | -34.361 [-59.73 to -9.38] | -42.653 [-61.39 to -17.29] | 21.053 [8.00 to 54.55] | -17.891 [-27.39 to 12.52]
Statistical Analysis 1: Comparison: Placebo vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.142, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Denosumab 210 mg Q6M; Test type: Superiority or Other; p = 0.218, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Denosumab 100 mg Q6M; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.010, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Denosumab 14 mg Q6M; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Denosumab 30 mg Q3M; Test type: Superiority or Other; p = 0.010, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Denosumab 14 mg Q3M; Test type: Superiority or Other; p = 0.020, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Denosumab 6 mg Q3M; Test type: Superiority or Other; p = 0.020, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 48 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo | Denosumab 6 mg Q3M | Denosumab 14 mg Q3M | Denosumab 30 mg Q3M | Denosumab 14 mg Q6M | Denosumab 60 mg Q6M | Denosumab 100 mg Q6M | Denosumab 210 mg Q6M | Alendronate 70 mg
Serious Adverse Events (participants affected / at risk) | 5/46 | 7/43 | 13/44 | 9/40 | 7/53 | 5/47 | 9/41 | 6/46 | 8/46
Other Adverse Events (participants affected / at risk) | 43/46 | 38/43 | 39/44 | 35/40 | 44/53 | 42/47 | 38/41 | 41/46 | 42/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | Denosumab 6 mg Q3M (N=43) | Denosumab 14 mg Q3M (N=44) | Denosumab 30 mg Q3M (N=40) | Denosumab 14 mg Q6M (N=53) | Denosumab 60 mg Q6M (N=47) | Denosumab 100 mg Q6M (N=41) | Denosumab 210 mg Q6M (N=46) | Alendronate 70 mg (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gallbladder disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Follicle centre lymphoma, follicular grade I, II, III stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Bronchial hyperactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colostomy closure (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | Denosumab 6 mg Q3M (N=43) | Denosumab 14 mg Q3M (N=44) | Denosumab 30 mg Q3M (N=40) | Denosumab 14 mg Q6M (N=53) | Denosumab 60 mg Q6M (N=47) | Denosumab 100 mg Q6M (N=41) | Denosumab 210 mg Q6M (N=46) | Alendronate 70 mg (N=46)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 5
Palpitations (Cardiac disorders) | 0 | 1 | 2 | 1 | 3 | 1 | 0 | 0 | 1
Blepharitis (Eye disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 3 | 3 | 3 | 3 | 2 | 4 | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 1 | 4 | 3 | 2 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 1 | 2 | 1 | 3 | 3 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 3 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 3 | 2 | 2 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 5 | 5 | 3 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 5 | 3 | 3 | 1 | 6 | 5 | 4
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 5 | 5 | 1 | 12 | 6 | 6 | 4 | 12
Flatulence (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 2 | 3 | 0 | 3 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 3 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 8 | 2 | 5 | 8 | 8 | 4 | 5 | 7
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 3 | 6 | 6 | 6 | 5 | 3 | 9 | 10
Stomach discomfort (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
Toothache (Gastrointestinal disorders) | 1 | 3 | 0 | 1 | 1 | 2 | 0 | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2 | 3 | 1 | 1 | 1 | 2 | 2
Chills (General disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 3 | 2 | 1 | 4 | 2 | 1 | 4 | 2
Influenza like illness (General disorders) | 5 | 4 | 4 | 3 | 10 | 11 | 6 | 3 | 7
Injection site bruising (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0
Injection site erythema (General disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 5 | 0 | 1 | 4 | 2 | 4 | 1 | 3 | 3
Pain (General disorders) | 0 | 3 | 4 | 1 | 2 | 1 | 1 | 3 | 3
Hypersensitivity (Immune system disorders) | 1 | 2 | 0 | 0 | 1 | 3 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 2 | 3 | 2 | 4 | 3 | 3 | 0 | 2 | 1
Bronchitis (Infections and infestations) | 5 | 2 | 1 | 10 | 4 | 3 | 1 | 5 | 4
Dental caries (Infections and infestations) | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 3 | 1 | 0 | 2 | 1 | 1
Ear infection (Infections and infestations) | 1 | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 1 | 1 | 1 | 1 | 1 | 4 | 2 | 3
Herpes zoster (Infections and infestations) | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 3 | 0
Nasopharyngitis (Infections and infestations) | 7 | 11 | 9 | 4 | 4 | 11 | 11 | 10 | 6
Pneumonia (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 3 | 2 | 1 | 1
Sinusitis (Infections and infestations) | 9 | 4 | 2 | 6 | 10 | 6 | 7 | 2 | 6
Tooth infection (Infections and infestations) | 0 | 3 | 0 | 1 | 3 | 2 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 11 | 15 | 10 | 8 | 13 | 16 | 8 | 18 | 14
Urinary tract infection (Infections and infestations) | 2 | 3 | 4 | 8 | 5 | 6 | 5 | 8 | 6
Viral infection (Infections and infestations) | 0 | 3 | 1 | 1 | 4 | 3 | 1 | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 4 | 1 | 1 | 0 | 3 | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 2 | 1 | 6 | 5 | 4 | 6 | 6 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 5 | 1 | 5 | 4 | 1 | 3
Foot fracture (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 2 | 2 | 4 | 1 | 4 | 1
Joint sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 3 | 3 | 4 | 2 | 2 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 1 | 0 | 3 | 1 | 2 | 3
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 2 | 4 | 3 | 0 | 3 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 3 | 5 | 2 | 2 | 7 | 2 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 7 | 13 | 9 | 12 | 11 | 10 | 12 | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 2 | 2 | 1 | 3 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 8 | 13 | 5 | 10 | 8 | 10 | 9 | 7
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 2 | 3 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 2 | 1 | 0 | 2 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 0 | 4 | 1 | 2 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 4 | 4 | 3 | 6 | 5 | 5 | 5 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3 | 1 | 1 | 3 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 1 | 5 | 5 | 2 | 5 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 1 | 3 | 2 | 3 | 2 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 2 | 0 | 2 | 1 | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 6 | 6 | 7 | 11 | 7 | 5 | 13 | 7
Shoulder pain (Musculoskeletal and connective tissue disorders) | 7 | 6 | 5 | 2 | 3 | 6 | 6 | 2 | 4
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 2 | 0 | 2 | 4 | 2 | 2
Dizziness (Nervous system disorders) | 4 | 1 | 5 | 3 | 6 | 4 | 2 | 1 | 4
Headache (Nervous system disorders) | 8 | 1 | 6 | 3 | 9 | 6 | 5 | 8 | 5
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 2 | 0
Migraine (Nervous system disorders) | 1 | 0 | 1 | 1 | 4 | 3 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 2 | 1 | 4 | 1 | 2 | 1 | 2 | 0 | 0
Sciatica (Nervous system disorders) | 2 | 2 | 2 | 5 | 2 | 2 | 2 | 3 | 1
Anxiety (Psychiatric disorders) | 2 | 0 | 2 | 1 | 5 | 1 | 0 | 4 | 3
Depression (Psychiatric disorders) | 4 | 0 | 3 | 6 | 6 | 2 | 1 | 3 | 3
Insomnia (Psychiatric disorders) | 0 | 2 | 6 | 4 | 4 | 4 | 1 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 3 | 1 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 4 | 3 | 3 | 2 | 5 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 1 | 4 | 2 | 3 | 3 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 5 | 2 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 2 | 3 | 1 | 3 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 1 | 1 | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 1 | 1 | 2 | 0 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 4 | 3 | 2 | 3 | 5 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0 | 2 | 3 | 0 | 0 | 2
Hot flush (Vascular disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 3 | 3
Hypertension (Vascular disorders) | 2 | 4 | 8 | 5 | 12 | 5 | 10 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.